CLINICAL TRIAL: NCT00401882
Title: Treatment of Ventricular Tachyarrhythmias Refractory To Shock With Beta Blockers: The SHOCK and BLOCK Trial
Acronym: Shock n Block
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult accrual
Sponsor: David Haines, MD (Other)
Collaborators: Medtronic BRC (Industry)
Responsible Party: Sponsor-Investigator, David Haines, MD, Coordinator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-008
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-03

CONDITIONS: Cardiac Arrest; Sudden Cardiac Death; Ventricular Fibrillation; Tachycardia, Ventricular
Keywords: Cardiac arrest; Sudden Cardiac Death; Ventricular Fibrillation; Pulseless Ventricular Tachycardia; Cardiopulmonary resuscitation
MeSH Terms: conditions — Heart Arrest; Death, Sudden, Cardiac; Ventricular Fibrillation; Tachycardia, Ventricular | interventions — Epinephrine; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- Standard Of Care Drug Epinephrine (Active Comparator): Additional doses of Epinephrine (1 mg) given as part of standard of care during cardiac arrest
  Interventions: Drug: Epinephrine
- IV Metoprolol instead Epinephrine (Active Comparator): IV metoprolol 5 mg. up to 2 times (only) during cardiac arrest will be given instead of additional Epinephrine doses
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Epinephrine — Epinephrine (1 mg) IV additional doses
  Other Names: adrenaline
  Arms: Standard Of Care Drug Epinephrine
Drug: Metoprolol — Metoprolol 5 mg IV (up to two times only) instead of epinephrine additional doses
  Other Names: lopressor
  Arms: IV Metoprolol instead Epinephrine

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of metoprolol, a "beta blocker," in treating patients in the hospital with a cardiac arrest. It will be given intravenously (given into a vein). The subjects who will take part in this study are 18 years of age or older, are experiencing a cardiac arrest in the hospital, and are in a life threatening situation. Patients who develop a cardiac arrest require prompt electrical defibrillation (electrical shocks) to restore the normal beating rhythm of the heart. In patients who do not respond to electrical defibrillation, current standard of care recommends the use of medications which have been shown to be of unknown benefit. Some people recover from a cardiac arrest, but many people do not. We want to learn whether giving metoprolol will improve survival of patients with a cardiac arrest. A total of 100 patients will be enrolled in the study. Patients will receive either the standard of care with the drug epinephrine or the standard of care plus metoprolol.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) is a catastrophic event and most commonly results from acute ventricular tachyarrhythmias (abnormal and lethal heart rhythms). It is often triggered by acute coronary events, which may occur in persons without known cardiac disease or in association with structural heart disease. Advanced therapies such as thrombolytic agents, percutaneous coronary intervention, and implantable cardioverter defibrillators are of no value to thousands of victims who do not survive. Many instances of SCD cannot be predicted and any intervention directed toward the general population would have to be applied to an estimated 1000 persons for every 1 person in whom SCD might be prevented. Thus, it would be reasonable to develop new treatment strategies to improve response to resuscitative efforts.

Prompt electrical defibrillation (electrical shocks) is the treatment of choice in persons who develop SCD due to ventricular fibrillation (VF) or pulseless ventricular tachycardia (pVT). However, in up to 25% of all cardiac arrests, patients develop shock resistant VF, defined as VF persisting beyond three defibrillation attempts, and 87-97% of these patients die. Medical therapy, including antiarrhythmic agents, sympathomimetic agents (i.e. stimulants), and buffers have been relegated to a secondary role since there is little evidence that they are of benefit and there use is considered indeterminate or class IIB. Furthermore, the "Guidelines 2000 for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care" of the American Heart Association and the International Liaison Committee on Resuscitation recommend antiarrhythmic drugs as "acceptable" and "probably helpful" in the treatment of VF that persists after three or more external defibrillation shocks. It has been previously reported that the survival rate of hospital patients suffering a cardiac arrest in which epinephrine was required was only 6%. Furthermore, Dorian et al reported a survival to hospital admission of 22.8% in patients suffering an out of hospital cardiac arrest and receiving amiodarone. It is believed that the acute effects of amiodarone are due to the class II or beta blocking effects of the drug.

Resuscitation can only be considered successful if the survivor has no disabling cognitive function. The American Heart Association/International Liaison Committee on Resuscitation guidelines state that with a duration of cardiac arrest of > 8 to 10 minutes, the frequency of significant, permanent neurologic damage becomes unacceptably high. Newer treatment modalities are needed to improve patient outcomes.

Epinephrine has been used during cardiopulmonary resuscitation for more than 100 years yet its use has become controversial because it is associated with increased myocardial oxygen consumption, ventricular tachyarrhythmias, and myocardial dysfunction during the period after resuscitation. The current International Guidelines on Emergency Cardiac Care cite both epinephrine and vasopressin as acceptable vasopressor drugs for treatment of refractory VF but neither drug is acknowledged to be of proven benefit.

Beta blockers might improve patient outcomes by blunting the adverse affects of a hyperadrenergic state that occurs during a cardiac arrest and by improving the balance between myocardial oxygen supply and demand. Ditchey et al showed in an animal model that pretreatment with a beta blocker prior to cardiac arrest followed by standard epinephrine therapy results in reduced myocardial injury during CPR without compromising successful defibrillation or post resuscitation left ventricular function.

The current research protocol was formulated in an attempt to develop new treatment options for patients who develop an in-hospital VF or pVT arrest refractory to electrical defibrillation with the specific goal of improving patient outcomes. The trial will utilize pre-filled, blinded syringes of Metoprolol in patients who develop an in-hospital cardiac arrest due to ventricular fibrillation or pulseless ventricular tachycardia (see study protocol).

Sudden cardiac death (SCD) claims approximately 250,000 persons annually in the United States. Ventricular fibrillation (VF) or pulseless ventricular tachycardia (pVT) appear to be responsible for 25-35% of all out of hospital episodes of sudden cardiac death. The reported average survival to hospital discharge following in-hospital arrest is just as poor at approximately 14-17% despite the development of widespread implementation of basic and advanced cardiac life support. Current American Heart Association (AHA) guidelines recommend prompt electrical defibrillation to reestablish organized electrical activity. Increasing duration of VF (i.e. "shock resistant VF") can result in two major adverse effects. First, an increased duration can reduce the ability to terminate the arrhythmia8. Second, if VF continues for more than four minutes, there is irreversible damage to the central nervous system and other organs. Despite aggressive efforts, successful resuscitation from out-of-hospital cardiac arrest occurs in only one third of patients and only about 10% of all patients are ultimately discharged from the hospital, many of whom are neurologically impaired. Also, the outcome of patients who suffer an in-hospital cardiac arrest is poor with reported survival to hospital discharge rates of 10-15%. Thus, despite improvements and advances in the treatment of heart disease, the outcome of patients experiencing SCD remains poor.

Prompt and early defibrillation of VF or pVT has become the standard of care. Drug therapy for shock resistant VF or pVT has been relegated to a secondary role since there is little evidence that these agents are of benefit. As a result, their use is considered indeterminate or class IIB. In addition, cardiac arrest and cardiopulmonary resuscitation are extreme forms of stress that lead to the highest catecholamine levels ever recorded in both human or experimental animal models. Endogenous catecholamine concentrations are high during ventricular fibrillation even in the absence of epinephrine administration. Currently, epinephrine is the vasopressor of choice for the treatment of cardiac arrest although vasopressin has been used as an alternative. Of note, vasopressin has been shown to be superior to epinephrine in patients with asystole however, its effects were similar to those of epinephrine in the management of VF or pulseless electrical activity. Furthermore, previous studies have raised concern that epinephrine's beta adrenergic effect may increase the myocardial oxygen consumption of the fibrillating heart and predispose to post-defibrillation dysfunction and cardiac arrhythmias.

Numerous animal studies have shown that beta adrenergic blockade reduces myocardial injury and improves survival. Kudenchuk, et al undertook a study in patients with out of hospital cardiac arrest due to ventricular fibrillation. Patients were randomized to receive either amiodarone or placebo after three consecutive defibrillations and one dose of epinephrine. The authors concluded that patients who received amiodarone had a higher rate of survival to hospital admission. It is felt that the beneficial effects are related to the initial class II or beta blocking properties of amiodarone. Furthermore, Dorian, et al reported a higher rate of survival to hospital admission in patients who received amiodarone as compared to lidocaine for shock resistant out-of-hospital ventricular fibrillation. Analysis from the European Myocardial Infarct Amiodarone Trial and the Canadian Amiodarone Myocardial Infarction Trial revealed an interaction between beta-blockers and amiodarone, specifically, the combination group had a better survival and the interaction was statistically significant for arrhythmic death or resuscitated arrest.

ELIGIBILITY:
Inclusion Criteria:

* All patients age > 18 years of age who develop an in-hospital VF or pVT arrest which persists after three or more precordial shocks.
* Patients who develop an in-hospital cardiac arrest due to asystole or PEA which subsequently converts to VF or pVT will be included.

Exclusion Criteria:

* Pediatric patients
* Pregnancy
* Age < 18 years of age
* Patients who develop VF or pVT in the emergency room, operating room or surgical intensive care unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-01; Primary Completion 2011-06 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Haines, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients in the ventricular tacchycardia refractory to shock with beta blocker
Pre-assignment Details: After the patient was refractory to treatment of the Epinephrine the patient would receive medication called Metroprolol
Groups:
- Additional Doses of Epinephrine: Epinephrine: additional doses Epinephrine (1 mg) IV given as part of standard of care in cardiac arrest
- Metoprolol Instead of Additional Epinephrine Doses: Metoprolol: Metoprolol 5 mg IV (up to two times) instead of additional doses of epinephrine
Period: Overall Study
Arm/Group | Additional Doses of Epinephrine | Metoprolol Instead of Additional Epinephrine Doses
Started | 2 | 5
Completed | 2 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Additional Epinephrine Doses: Additional Epinephrine (1 mg) IV doses as part of standard of care in cardiac arrest
- Metoprolol: Metoprolol 5 mg IV (up to two doses only) instead of additional epinephrine doses in cardiac arrest
- Total: Total of all reporting groups
Arm/Group | Additional Epinephrine Doses | Metoprolol | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (21.9) | 60.8 (5.49) | 63 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Return of Spontaneous Circulation
Description: The patient will be evaluated for sufficiently stable and organized rhythm and blood pressure.
Time Frame: After electrical defibrillation
Measure: Count of Participants; unit: Participants
Groups:
- Additional Doses of Epinephrine: Epinephrine: Additional doses of epinephrine (1 mg IV) given as part of standard of care during cardiac arrest
- Metoprolol Instead of Additional Epinephrine Doses: Metoprolol 5 mg IV (up to 2 times) instead of additional epinephrine doses
Arm/Group | Additional Doses of Epinephrine | Metoprolol Instead of Additional Epinephrine Doses
Number analyzed (Participants) | 2 | 5
Participants | 0 | 1

2. Secondary Outcome: Survival to Hospital Discharge
Description: the number of patients who are alive at hospital discharge
Time Frame: from time of arrest to discharge or death
Measure: Count of Participants; unit: Participants
Groups:
- Additional Epinephrine Doses: Additional doses of Epinephrine (1 mg) given as part of standard of care during cardiac arrest
  Epinephrine: Epinephrine (1 mg) IV additional doses
- Metoprolol Instead of Additional Epinephrine Doses: IV metoprolol 5 mg. (up to 2 times only) during cardiac arrest will be given instead of additional Epinephrine doses
  Metoprolol: Metoprolol 5 mg IV (up to two times only) instead of epinephrine additional doses
Arm/Group | Additional Epinephrine Doses | Metoprolol Instead of Additional Epinephrine Doses
Number analyzed (Participants) | 2 | 5
Participants | 0 | 0

3. Secondary Outcome: Adverse Effects
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Additional Doses of Epinephrine: Epinephrine: Additional doses of epinephrine IV (1 mg) given as part of standard of care in cardiac arrest
- Metoprolol Instead of Additional Epinephrine Doses: Metoprolol: Metoprolol 5mg IV (up to two times only) instead of additional epinephrine doses
Arm/Group | Additional Doses of Epinephrine | Metoprolol Instead of Additional Epinephrine Doses
Number analyzed (Participants) | 2 | 5
Participants | 0 | 0

4. Secondary Outcome: Number of Precordial Shocks Required After the Administration of Metoprolol or Epinephrine
Time Frame: 120 minutes
Population: Data point not analyzed
Arm/Group | Additional Epinephrine Doses | Metoprolol
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Total Duration of Resuscitative Efforts
Time Frame: 120 minutes
Population: Data point not analyzed
Arm/Group | Additional Epinephrine Doses | Metoprolol
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Need for Additional Antiarrhythmic Drugs
Time Frame: 120 minutes
Population: Data point not analyzed
Arm/Group | Additional Epinephrine Doses | Metoprolol
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: After Electrical Defibrillation, up to 30 days.
Groups:
- Additional Doses of Epinephrine: Epinephrine: Additional doses epinephrine (1 mg IV) as part of standard of care during cardiac arrest
- Metoprolol Instead of Additional Doses of Epinephrine: Metoprolol: Metoprolol 5 mg IV (up to two times) instead of additional epinephrine doses
Arm/Group | Additional Doses of Epinephrine | Metoprolol Instead of Additional Doses of Epinephrine
All-Cause Mortality (participants affected / at risk) | 2/2 | 5/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 0/2 | 0/5

LIMITATIONS AND CAVEATS:
Early termination secondary to poor enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No